CLINICAL TRIAL: NCT03339674
Title: Sub-Project No 8 of the Research Group RISKDYNAMICS: Addiction Risk - the Dynamic of Risk Perception and Risk Behavior in Alcohol Dependence, Work Package 1, Study 1.
Brief Title: Addiction Risk: Psychoeducational Intervention to Change Risk Perception Among Alcohol Patients in Residential Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Centre for Psychiatry Reichenau, Germany (Unknown)
Responsible Party: Principal Investigator, Michael Odenwald, Director Psychotherapy Outpatient Clinic, University of Konstanz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OD 113/2-1
Record Dates: First submitted 2017-05-10; First posted 2017-11-13 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Psychoeducational Group Intervention on Alcohol Drinking Related to Stress: Psychological group intervention with 3 sessions of 60 min (Odenwald & Semrau, 2012). Contains psychoeducation on alcohol drinking related to stress and PTSD.
  Interventions: Behavioral: Psychoeducational Group Intervention on Alcohol Drinking Related to Stress
- Control (Active Comparator): Cognitive Training: Psychological group intervention with 3 sessions of 60 min. The content is paper-and-pencil based cognitive training of memory and attention functions.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Psychoeducational Group Intervention on Alcohol Drinking Related to Stress — Manualized and standardized psychotherapeutic group intervention with three sessions of 60 min duration each which are to be delivered in a one-week period.
  Arms: Intervention
Behavioral: Cognitive Training — Manualized and standardized psychotherapeutic group intervention with three sessions of 60 min duration each which are to be delivered in a one-week period.
  Arms: Control

SUMMARY:
Based on previous research (Odenwald & Semrau, 2012) the investigators know that psychoeducation on comorbid mental disorders during residential alcohol detoxification can improve subsequent treatment utilization. In this study they will study a hypothesized psychological mechanism that contributes to this behavior change.

The investigators will recruit alcohol dependent patients in residential detox treatment who all receive Treatment as Usual. Participants will be randomly assigned to an additional psychoeducational group therapy (intervention group) or to an additional neuropsychological group training (control group). Measurements will take place on the day before study inclusion, one week later and one month after release from index residential treatment. Measurements will include alcohol-related risk perception, alcohol use, treatment motivation, comorbid psychiatric symptoms and whether the patient has regularly completed treatment and whether he/she has been transferred to subsequent treatment. Furthermore, six months after release from index treatment information on re-admission to the clinic is assessed from patient files.

The investigators hypothesize that the behavioral effects of psychoeducational group intervention will be mediated by adaptive changes of the individual's alcohol-related risk perception.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependence (according to ICD-10)

Exclusion Criteria:

* treatment episode is acute crisis intervention
* acute psychosis
* acute suicidality
* no command of German language (reading writing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Alcohol-related Risk Perception | one week
  The patient's self-reported rating of the patient's own perception of alcohol-related risks in the German Questionnaire on Alcohol-related Risk Perception (Klepper, Odenwald & Rockstroh, 2016).

SECONDARY OUTCOMES:
Treatment completion | One month after study completion
  Binary variable: The patient regularly completes the residential detox treatment or he/she can prematurely end the treatment (treatment drop out).
Transfer to subsequent treatment | One month after study completion
  Binary variable: Patient is directly transferred from detox treatment unit to subsequent alcohol in-patient or day-clinic treatment.
Alcohol relapse | four weeks
  Drinking alcohol after treatment
Readmission to detox treatment | six months
  The patient is readmitted to the same alcohol detox treatment unit

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Psychiatry Reichenau, Reichenau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odenwald M, Semrau P. Reducing dropout among traumatized alcohol patients in detoxification treatment: a pilot intervention study. Eur Addict Res. 2012;18(2):54-63. doi: 10.1159/000333336. Epub 2011 Dec 16. PMID 22178762